CLINICAL TRIAL: NCT00350467
Title: A Randomized, 6-week Double-blind, Parallel Study to Evaluate the Efficacy and the Safety of Flexible Doses of Extended Release OROS Paliperidone Compared With Olanzapine in the Treatment of Patients With Schizophrenia
Brief Title: A Randomized, Active-controlled, Double-blind, Parallel-Goup Study of the Efficacy and Safety of Extended Release(ER) Paliperidone in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR010861
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-05

CONDITIONS: Acute Schizophrenia
Keywords: Schizophrenia; DSM-IV; PANSS; informed consent
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

INTERVENTIONS:
Drug: ER OROS paliperidone and Olanzapine

SUMMARY:
This is a randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), active-controlled, flexible-dose, parallel group, multicenter study. The study consists of a screening phase, a double-blind treatment phase (6 weeks) and a safety follow-up phase (1 week).

The patients in this study will be randomized to 1 of 2 treatment groups to receive extended release OROS paliperidone or Olanzapine once daily for the 6-week double-blind treatment phase. Randomization will occur in a ratio of 1 (extended release OROS paliperidone) to 1 (Olanzapine). Patients must be hospitalized at least 14 days after entry. Those who receive extended release OROS paliperidone will start at a dosage of 6 mg taken daily, dose may be titrated up by 3mg/day every 7 days, or down rapidly based on the balance of efficacy (effectiveness of drug) and safety/tolerability assessed by the investigator. After the initial 7 days, dose could be flexible within 3-12mg/day. Those who receive olanzapine will start at a dosage of 5mg taken daily, dose may be titrated up by 5mg/day every 7 days, or down rapidly based on the balance of efficacy and safety/tolerability assessed by the investigator. After the initial 7 days, dose could be flexible within 5-15mg/day.

Efficacy parameters include Positive and Negative Symptom Scale (PANSS) score, Clinical Global Impression-Severity (CGI-S) and Personal and Social Performance (PSP) score per assessment visit. The primary efficacy is the change in PANSS from baseline to the last post-randomization assessment. Safety assessments include the adverse events, changes in physical examination, vital signs, laboratory tests at pretreatment and posttreatment.

DETAILED DESCRIPTION:
The study hypothesis is that the effect of extended release OROS paliperidone is not worse than that of Olanzapine in the treatment of schizophrenia as measured by the change in PANSS from baseline to the last post-randomization assessment. A flexible dose range is used in this study. The flexible dose of paliperidone is ranged from 3 to 12mg/day. The flexible dose of olanzapine is ranged from 5-15mg/day.The study medication is capsulized to maintain blind. Study medication must be taken orally once daily before 10 AM with or without food in a consistent manner throughout the study. Medication can not be chewed, divided, dissolved, or crushed. Treatment duration is 6 week each subject.

ELIGIBILITY:
Inclusion Criteria:

* Patients (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* DSM-IV diagnosis of schizophrenia (295.10, 295.20, 295.30, 295.60, 295.90) at entry
* Total PANSS score at screening and baseline between 60 and 120, inclusive
* Female patients must be postmenopausal for at least 1 year, surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch) before entry (and agree to continue that method throughout the study) - abstinence is not an acceptable method
* have a negative urine b hCG pregnancy test at screening
* Capable of self-administering study drug, or has consistent help and support available throughout the study to do this

Exclusion Criteria:

* A DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) Axis I diagnosis other than schizophrenia
* Inability to swallow the study drug whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drug, as this may affect the release profile)
* Previous history of a lack of response to any antipsychotic (lack of response defined as subject having had least twice a documented medical history of no clinical response despite adequate doses and durations of treatment, or the inability to tolerate effective doses)
* Significant risk of suicidal or violent behavior
* Injection of a depot antipsychotic within 120 days before screening, or use of paliperidone palmitate within 10 months before screening
* Use of monoamine oxidase inhibitors within 4 weeks before screening
* Use of antidepressants other than monoamine oxidase inhibitors or mood stabilizers (e.g., antiepileptics, lithium) within 2 weeks before screening
* Received electroconvulsive therapy within 3 months before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2006-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in total PANSS score at endpoint (6-week double-blind or last assessment after baseline) from baseline.

SECONDARY OUTCOMES:
Changes in PANSS positive and negative scores at each assessment time point from baseline; Changes in CGI-S at each assessment time point from baseline; Changes in PSP at each assessment time point from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd. Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (7):
- China (7):
  - Beijing, Beijing Municipality
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Nanjing, Jiangsu
  - Shanghai, Shanghai Municipality
  - Suzhou, Zhejiang
  - Xi'an

REFERENCES:
- [Background] Fowler JA, Bettinger TL, Argo TR. Paliperidone extended-release tablets for the acute and maintenance treatment of schizophrenia. Clin Ther. 2008 Feb;30(2):231-48. doi: 10.1016/j.clinthera.2008.02.011. PMID 18343262
- See also: A Randomized, 6-Week Double Blind, Parallel Study to Evaluate the Efficacy and the Safety of Flexible Doses of Extended Release OROS Paliperidone Compared with Olanzapine in the Treatment of Patients With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1078&filename=CR010861_CSR.pdf